CLINICAL TRIAL: NCT03086200
Title: CCTG 603: Randomized Controlled Trial of iTAB Plus Motivational Interviewing for PrEP Adherence in Transgender Individuals (The iM-PrEPT Study)
Brief Title: Randomized Controlled Trial of iTAB Plus Motivational Interviewing for PrEP Adherence in Transgender Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Southern California (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Los Angeles LGBT Center (Other); Family Health Centers of San Diego (Other)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCTG 603
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Patient Adherence; HIV Seronegativity
Keywords: PrEP; Pre-exposure Prophylaxis; Text messaging; Truvada; Motivational interviewing; Transgender; Gender Non-conforming
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- iTAB + SOC Control Arm (No Intervention): Participants will receive PrEP and standard of care (SOC) including health education, clinical assessments, laboratory safety monitoring, STI and HIV screening, HIV risk reduction counseling, assessment of psychosocial barriers, and adherence counseling. In addition to SOC, participants will receive daily text messages (iTAB) as reminders for medication adherence. Text messages will be setup during the Baseline visit in coordination with the participant's preferences.
- iTAB + MI-b Intervention Arm (Experimental): Participants will receive the same PrEP, SOC procedures, and iTAB support as that of the Control Arm. Participants in the Intervention Arm will also receive brief motivational interviewing counseling sessions if adherence becomes suboptimal. Adherence will be monitored by responses to the iTAB system; if Intervention Arm participants reply with 3 consecutive negative or non-responses, MI-b counselors will perform 15-minute over-the-phone motivational interviewing counseling sessions with the participant.
  Interventions: Behavioral: brief Motivational Interviewing

INTERVENTIONS:
Behavioral: brief Motivational Interviewing — All study participants will receive daily dosing text message reminders.
  Participants randomized to the MI-b Intervention and who are persistently non-adherence based on negative or non-responses to iTAB will be sent automated high alert messages notifying the participant to take their study medication and respond to iTAB. Both the study coordinator and the MI counselor will also receive the high alert message. Participants will be contacted by the MI counselor for a phone MI-b session within 72 hours of a high alert message to discuss adherence. Participants who continue to be non-adherent despite receiving these messages will be switched to receive alert messages on a monthly schedule.
  Arms: iTAB + MI-b Intervention Arm

SUMMARY:
CCTG 603 is an open-label, two-arm, randomized (1:1) clinical demonstration project to determine if brief Motivational Interviewing (MI-B) added to a text-message based adherence intervention (iTAB) improves adherence to PrEP among transgender persons.

DETAILED DESCRIPTION:
A total of 300 HIV-uninfected transgender or gender non-conforming individuals, defined as currently identifying as a gender different from sex assigned at birth, with high-risk transmission behavior will be enrolled into this study. Each participant will be followed for a maximum of 48 weeks after enrollment. The primary endpoint will be measured at 48 weeks, or the last week on study if the participant is discontinued early.

All participants will start PrEP with TDF / FTC fixed dose combination taken once daily. Subjects will be randomized (1:1) to the iTAB text messaging adherence reminder intervention either with or without brief motivational interviewing (MI-b) for suboptimal adherence. All participants will receive the iTAB system to provide personalized, automated text messages to support and monitor adherence. In the MI-b arm, poor adheres by iTAB reporting will receive targeted MI-b via telephone.

Both groups will receive PrEP in accordance with standardized comprehensive methods of prescribing, which includes risk reduction counseling, adherence counseling, and clinical assessments with safety monitoring, as well as HIV and STI screening.

ELIGIBILITY:
Inclusion Criteria:

* Transgender identity, defined as identifying differently from sex assigned at birth
* Age 18 years or older
* Risk of acquisition of HIV as evident by one or more of the following:

Has at least one HIV infected sexual partner for ≥4 weeks

OR,

Anticipated or concern of unprotected anal or vaginal sex with a partner in the next 3 months

OR,

Any partner in the past 12 months AND at least one of the following:

1. any condomless anal or vaginal sex in the past 12 months
2. any STI diagnosed or reported in the past 12 months
3. exchange of money, gifts, shelter, or drugs for sex

OR,

PEP-use in the past 12 months

* Negative for HIV infection by nucleic acid test (NAT) or other sensitive method such as 4th generation antigen/antibody test
* Acceptable renal function as measured by calculated creatinine clearance of at least 60 mL/min by the Cockcroft-Gault formula (eCcr (male) in mL/min = [(140 - age in years) x (lean body weight in kg)] / (72 x serum creatinine in mg/dL) in the past 30 days

Exclusion Criteria:

* Unable to give informed consent
* Active hepatitis B defined by a positive hepatitis B surface antigen (HBsAg)
* Substantial medical condition that, in the opinion of the investigator, would preclude participation, as defined by

  * gastrointestinal condition that would impair absorption of study drugs
  * known condition of reduce bone density (e.g. osteoporosis or osteogenesis imperfect) that significantly elevate the risk of bone fracture
  * neurological or severe psychiatric condition that would significantly impair the ability to adhere to PrEP
  * tubular or glomerular kidney disease that could be exacerbated by tenofovir
  * other medical condition that would unacceptably increase the risk of harm from study drug or significantly impair the ability to adhere to PrEP
* Suspected sensitivity or allergy to the study drug or any of its components
* Currently using an essential product or medication that interacts with the study drug such as the following:

  * other antiretroviral agent (including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, integrase inhibitors, protease inhibitors or investigational antiretroviral agents) - if currently on TDF/FTC for PEP or PrEP they can switch to study provided drug but can not continue any other antiretroviral agent
  * agents with known nephrotoxic potential:
  * aminoglycoside antibiotics (including gentamicin)
  * IV amphotericin B
  * cidofovir
  * cisplatin
  * foscarnet
  * IV pentamidine
  * IV vancomycin
  * oral or IV gancyclovir
  * other agents with significant nephrotoxic potential
  * drugs that slow renal excretion
  * probenecid
  * immune system modulators
  * systemic chemotherapeutic agents (i.e. cancer treatment medications)
  * ongoing systemic corticosteroids (with the exception of short courses of tapering steroid doses for asthma or other self- limited condition).
  * interleukin-2 (IL-2)
  * interferon (alpha, beta, or gamma)
  * other agent known to have a significant interaction with TDF or FTC
* Proteinuria 2+ or greater by urine dipstick
* Pregnancy (if individual has a uterus)
* Other condition that, in the opinion of the investigator, would put the participant at risk, complicate interpretation of study outcome data, or would otherwise interfere with participation or achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender or Gender Non-conforming, defined as identifying with a gender different from sex assigned at birth.
Enrollment: 263 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
PrEP Adherence | Baseline up to Week 48
  To compare adherence to fixed dose TDF/FTC, as measured by intracellular levels of TFV-DP > 1246 fmol/punch, between subjects randomized to receive iTAB with versus without brief Motivational Interviewing, when used for adherence support to pre-exposure prophylaxis among transgender individuals at elevated risk for HIV acquisition.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Morris, MD MPH, Principal Investigator — CCTG, UCSD AVRC; David Moore, PhD, Study Chair — CCTG, UCSD HNRP
Locations (5):
- United States (5):
  - Los Angeles Lesbian, Gay, Bisexual, and Transgender Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Family Health Centers of San Diego, San Diego, California
  - University of California, San Diego, San Diego, California
  - LA Biomed at Harbor-UCLA, Torrance, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03086200/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03086200/ICF_001.pdf